CLINICAL TRIAL: NCT06840392
Title: A Randomized, Double-blind, Double-dummy, Placebo-controlled, Multicenter, Phase 3 Study Assessing the Efficacy, Safety, and Tolerability of 2 Doses of Remibrutinib Over a 68-week Treatment Period in Adult and Adolescent Patients With Moderate to Severe Hidradenitis Suppurativa (RECHARGE-2)
Brief Title: A Phase 3 Study to Assess Efficacy Safety and Tolerability of Remibrutinib in Adult and Adolescent Patients With Moderate to Severe Hidradenitis Suppurativa
Acronym: RECHARGE-2
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CLOU064J12302; 2024-513266-19-00 (Registry Identifier: EU CT Number)
Record Dates: First submitted 2025-02-17; First posted 2025-02-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Hidradenitis Suppurativa
Keywords: Bruton's tyrosine kinase (BTK) inhibitor; Hidradenitis Suppurativa; HS; Hidradenitis Suppurativa clinical response; HiSCR; remibrutinib; LOU064; Hidradenitides, Suppurativa; Hidradenitis, Suppurativa; Suppurativa Hidradenitides; Suppurativa Hidradenitis; Acne inversa,; Verneuil disease; Inflammatory skin disease; Chronic skin condition
MeSH Terms: conditions — Hidradenitis Suppurativa; Hidradenitis; Dermatitis | interventions — remibrutinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Remibrutinib Dose A (Treatment Period 1 and 2) (Experimental): articipants randomized to receive remibrutinib Dose A during Treatment Period 1 and 2
  Interventions: Drug: Remibrutinib Dose A
- Remibrutinib Dose B (Treatment Period 1 and 2) (Experimental): Participants randomized to receive remibrutinib Dose B during Treatment Period 1 and 2
  Interventions: Drug: Remibrutinib Dose B
- Placebo (Treatment Period 1) + remibrutinib Dose B (Treatment Period 2) (Placebo Comparator): Participants randomized to receive placebo during Treatment Period 1 followed by remibrutinib dose B during Treatment Period 2
  Interventions: Drug: Remibrutinib Dose B; Drug: Placebo 1; Drug: Placebo 2

INTERVENTIONS:
Drug: Remibrutinib Dose A — Remibrutinib Dose A (oral)
  Other Names: LOU064
  Arms: Remibrutinib Dose A (Treatment Period 1 and 2)
Drug: Remibrutinib Dose B — Remibrutinib Dose B (oral)
  Other Names: LOU064
  Arms: Placebo (Treatment Period 1) + remibrutinib Dose B (Treatment Period 2); Remibrutinib Dose B (Treatment Period 1 and 2)
Drug: Placebo 1 — Placebo matching to remibrutinib Dose A (oral)
  Arms: Placebo (Treatment Period 1) + remibrutinib Dose B (Treatment Period 2)
Drug: Placebo 2 — Placebo matching to remibrutinib Dose B (oral)
  Arms: Placebo (Treatment Period 1) + remibrutinib Dose B (Treatment Period 2)

SUMMARY:
The purpose of this study is to establish the efficacy, safety, and tolerability of remibrutinib (LOU064) Dose A and Dose B compared to placebo in participants with moderate to severe hidradenitis suppurativa (HS).

DETAILED DESCRIPTION:
The total duration of the study is 76 weeks and consists of: Screening (up to 4 weeks), Treatment Period 1 (16 weeks, double-blind treatment with remibrutinib (Dose A or Dose B) or placebo, Treatment Period 2 (52 weeks, treatment with remibrutinib (Dose A or Dose B) and Safety Follow-Up (treatment-free follow-up for 4 weeks).

Participants who prematurely discontinue study treatment (either during Treatment Period 1 or Treatment Period 2) are encouraged to remain in the study. Participants who do not wish to remain in the study will enter a 4-week Safety Follow-Up period.

ELIGIBILITY:
Key Inclusion Criteria:

1. Male and female participants ≥ 12 years of age at the time of signing of the informed consent.
2. Diagnosis of HS based on clinical history and physical examination for at least 6 months prior to the Baseline visit.
3. Participants with moderate to severe HS defined as:

   * A total of at least 5 AN count (abscesses and/or inflammatory nodules) AND
   * Inflammatory lesions should affect at least 2 distinct anatomic areas (e.g., left and right axillae)

Key Exclusion Criteria:

1. Presence of more than 20 fistulae/tunnels (both draining and non-draining) in total at baseline.
2. Any active skin disease or conditions that may interfere with the assessment of HS.
3. Previous exposure to remibrutinib or other BTK inhibitors.
4. Use of other investigational drugs within 5 half-lives of enrollment, or within 30 days (for small molecules) prior to randomization, or until the pharmacodynamic effect has returned to baseline (for biologics), whichever is longer.
5. Significant bleeding risk or coagulation disorders.
6. History of gastrointestinal bleeding.
7. Requirement for anti-platelet (except for acetylsalicylic acid up to 100 mg/d or clopidogrel up to 75 mg/d) or anti-coagulant medication.
8. History or current hepatic disease.
9. Evidence of clinically significant cardiovascular, neurological, psychiatric, pulmonary, renal, hepatic, endocrine, metabolic, hematological disorders, gastrointestinal disease or immunodeficiency that, in the Investigator's opinion, would compromise the safety of the participant, interfere with the interpretation of the study results or otherwise preclude participation or protocol adherence of the participant.
10. History of hypersensitivity to any of the study drug constituents.
11. Known or suspected infectious disease that is active, chronic or recurrent which precludes the participant from participating in the trial as per investigator's assessment. These infectious diseases include and are not limited to opportunistic infections (e.g., tuberculosis, atypical mycobacterioses, listeriosis or aspergillosis) and/or known or suspected Human Immunodeficiency Virus (HIV) infection. Should it be required by local regulations and/or considered appropriate by the investigator, an HIV test can be performed to confirm eligibility.
12. History of live attenuated vaccine administration within 6 weeks prior to randomization or requirement to receive these vaccinations at any time while on study treatment.
13. Major surgery within 8 weeks prior to screening or planned surgery for the duration of the study.

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 12 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 555 (Estimated)
Dates: Start 2025-03-20 (Actual); Primary Completion 2027-10-29 (Estimated); Study Completion 2028-03-17 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants with Hidradenitis Suppurativa clinical response 50 (HiSCR50) at Week 16 | Week 16
  HiSCR50 is defined as at least a 50% decrease in Abscess and Inflammatory Nodule (AN) count with no increase in the number of abscesses and in the number of draining tunnels/fistulae compared to baseline.

SECONDARY OUTCOMES:
Proportion of participants with Abscesses and inflammatory nodules 50 (AN50) response at Week 16 | Week 16
  AN50 is defined as at least a 50% decrease in Abscess and Inflammatory Nodule (AN) count compared to baseline
Percentage change from baseline in International Hidradenitis Suppurativa Severity Score System (IHS4) at Week 16 | From baseline up to Week 16
  The IHS4 is a disease severity scoring system developed by the European Hidradenitis Suppurativa Foundation. It is a weighted sum of different types of inflammatory lesion counts, calculated as 1 x number of nodules + 2 x number of abscesses + 4 x number of draining tunnels (=fistulae=sinuses).
Proportion of participants with HiSCR75 response at Week 16 | Week 16
  HiSCR75 is defined as at least a 75% decrease in Abscess and Inflammatory Nodule (AN) count with no increase in the number of abscesses and in the number of draining tunnels/fistulae compared to baseline.
Proportion of participants experiencing Hidradenitis Suppurativa (HS) flares at Week 16 | Up to Week 16
  Flare is defined as at least a 25% increase in AN count with a minimum increase of 2 AN relative to baseline.
Proportion of participants with HiSCR50 response at Week 8 | Week 8
  HiSCR50 is defined as at least a 50% decrease in Abscess and Inflammatory Nodule (AN) count with no increase in the number of abscesses and in the number of draining tunnels/fistulae compared to baseline.
Proportion of participants with HiSCR90 response at Week 16 | Week 16
  HiSCR90 is defined as at least a 90% decrease in Abscess and Inflammatory Nodule (AN) count with no increase in the number of abscesses and in the number of draining tunnels/fistulae compared to baseline.
Proportion of participants with clinical response in HS related skin pain (NRS 30), at worst at Week 16 | Week 16
  Achievement of NRS30 at Week 16, among participants with baseline NRS ≥ 3 (pooled data from studies CLOU064J12301 and CLOU064J12302).
  NRS30 is defined as at least a 30% reduction and at least 2-unit reduction from baseline in Patient's Global Assessment of Skin Pain - at worst over the past 7 days.
Incidence of treatment emergent adverse events and serious adverse events during the study | From randomization to end of study, assessed up to 72 weeks.
  The distribution of adverse events will be done via the analysis of frequencies for treatment emergent Adverse Event (TEAEs), Serious Adverse Event (TESAEs) and Deaths due to AEs, through the monitoring of relevant clinical and laboratory safety parameters.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (124):
- United States (36):
  - Total Skin and Beauty Dermatology Center PC, Birmingham, Alabama
  - CTT Research, Gilbert, Arizona
  - Ctr Dermatology and Plastic Surgery, Scottsdale, Arizona
  - Ctr for Dermatology Clinical Res, Fremont, California
  - USC Keck School of Medicine, Los Angeles, California
  - MedDerm Associates, San Diego, California
  - Driven Research, Coral Gables, Florida
  - Floridian Research Institute, Miami, Florida
  - Sarasota Arthritis Res Ctr, Sarasota, Florida
  - University Of South Florida, Tampa, Florida
  - Emory School of Med Dermatology, Atlanta, Georgia
  - Atlanta Biomedical Clin Res LLC, Atlanta, Georgia
  - Northwestern University, Chicago, Illinois
  - Endeavor Health, Glenview, Illinois
  - Dundee Dermatology, West Dundee, Illinois
  - Southern IN Clinical Trials, New Albany, Indiana
  - Beth Israel Deaconess Med Center, Boston, Massachusetts
  - Metro Boston Clinical Partners, Brighton, Massachusetts
  - Clinical Research Inst of MI, Chesterfield, Michigan
  - Deluxe Dermatology, St Louis, Missouri
  - Skin Specialists PC, Omaha, Nebraska
  - Vivida Dermatology, Las Vegas, Nevada
  - North Shore University Hospital, New Hyde Park, New York
  - Cameron Dermatology, New York, New York
  - Optima Research Boardman, Boardman, Ohio
  - Ohio State University, Columbus, Ohio
  - Wright State University, Fairborn, Ohio
  - Apex Clinical Research Center LLC, Mayfield Heights, Ohio
  - Clinical Research Ctr of Carolinas, Charleston, South Carolina
  - Goodlettsville Dermatology Research, Goodlettsville, Tennessee
  - Accurate Clinical Research, Humble, Texas
  - Austin Inst for Clinical Research, Pflugerville, Texas
  - Center for Clinical Studies-Lee, Webster, Texas
  - Care Access Alexandria, Arlington, Virginia
  - Complexions Dermatology, Danville, Virginia
  - Forefront Dermatology, Vienna, Virginia
- Argentina (4):
  - Novartis Investigative Site, Berazategui, Buenos Aires
  - Novartis Investigative Site, CABA
  - Novartis Investigative Site, Caba
  - Novartis Investigative Site, Córdoba
- Novartis Investigative Site, Linz, Austria
- Belgium (4):
  - Novartis Investigative Site, Brussels, Brussels Capital
  - Novartis Investigative Site, Woluwe-Saint-Lambert, Brussels Capital
  - Novartis Investigative Site, Leuven, Vlaams Brabant
  - Novartis Investigative Site, Liège
- Canada (5):
  - Novartis Investigative Site, Edmonton, Alberta
  - Novartis Investigative Site, London, Ontario
  - Novartis Investigative Site, Montreal, Quebec
  - Novartis Investigative Site, Québec, Quebec
  - Novartis Investigative Site, Sherbrooke, Quebec
- Colombia (3):
  - Novartis Investigative Site, Medellín, Antioquia
  - Novartis Investigative Site, Bogota, Cundinamarca
  - Novartis Investigative Site, Medellín
- Czechia (3):
  - Novartis Investigative Site, Karlovy Vary
  - Novartis Investigative Site, Plzen Bolevec
  - Novartis Investigative Site, Prague
- France (7):
  - Novartis Investigative Site, Brest
  - Novartis Investigative Site, La Rochelle
  - Novartis Investigative Site, Lyon
  - Novartis Investigative Site, Nice
  - Novartis Investigative Site, Reims
  - Novartis Investigative Site, Rouen
  - Novartis Investigative Site, Toulouse
- Germany (16):
  - Novartis Investigative Site, Freiburg im Breisgau, Baden-Wurttemberg
  - Novartis Investigative Site, Würzburg, Bavaria
  - Novartis Investigative Site, Frankfurt am Main, Hesse
  - Novartis Investigative Site, Düsseldorf, North Rhine-Westphalia
  - Novartis Investigative Site, Merzig, Saarland
  - Novartis Investigative Site, Leipzig, Saxony
  - Novartis Investigative Site, Bad Bentheim
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Dessau
  - Novartis Investigative Site, Dortmund
  - Novartis Investigative Site, Essen
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Lübeck
  - Novartis Investigative Site, Minden
  - Novartis Investigative Site, München
  - Novartis Investigative Site, Tübingen
- Greece (3):
  - Novartis Investigative Site, Athens
  - Novartis Investigative Site, Chaïdári
  - Novartis Investigative Site, Thessaloniki
- Hungary (6):
  - Novartis Investigative Site, Pécs, Baranya
  - Novartis Investigative Site, Debrecen, Hajdu Bihar Megye
  - Novartis Investigative Site, Debrecen, Hajdú-Bihar
  - Novartis Investigative Site, Budapest
  - Novartis Investigative Site, Kecskemét
  - Novartis Investigative Site, Szeged
- Malaysia (6):
  - Novartis Investigative Site, Kuala Lumpur, Kuala Lumpur
  - Novartis Investigative Site, Ipoh, Perak
  - Novartis Investigative Site, Kota Kinabalu, Sabah
  - Novartis Investigative Site, Johor Bahru
  - Novartis Investigative Site, Selangor Darul Ehsan
  - Novartis Investigative Site, Wilayah Persekutuan
- Novartis Investigative Site, Durango, Mexico
- Poland (2):
  - Novartis Investigative Site, Warsaw, Masovian Voivodeship
  - Novartis Investigative Site, Warsaw
- Alma Cruz-Santana Private Practice, Carolina, Puerto Rico
- Romania (3):
  - Novartis Investigative Site, Bucharest, District 2
  - Novartis Investigative Site, Bucharest
  - Novartis Investigative Site, Timișoara
- Spain (9):
  - Novartis Investigative Site, Granada, Andalusia
  - Novartis Investigative Site, Palma, Balearic Islands
  - Novartis Investigative Site, Barcelona
  - Novartis Investigative Site, Granollers
  - Novartis Investigative Site, Las Palmas GC
  - Novartis Investigative Site, Madrid
  - Novartis Investigative Site, Pontevedra
  - Novartis Investigative Site, Seville
  - Novartis Investigative Site, Valencia
- Turkey (Türkiye) (10):
  - Novartis Investigative Site, Izmir, Balcova
  - Novartis Investigative Site, Ankara, Bilkent-Cankaya
  - Novartis Investigative Site, Izmir, Buca
  - Novartis Investigative Site, Aydin, Efeler
  - Novartis Investigative Site, Denizli, Kinikli
  - Novartis Investigative Site, Ankara, Sihhiye-Altindag
  - Novartis Investigative Site, Ankara, Yenimahalle
  - Novartis Investigative Site, Mersin, Yenisehir
  - Novartis Investigative Site, Izmir
  - Novartis Investigative Site, Kecioren Ankara
- United Kingdom (4):
  - Novartis Investigative Site, Leeds, West Yorkshire
  - Novartis Investigative Site, Cardiff
  - Novartis Investigative Site, London
  - Novartis Investigative Site, Southampton

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com